CLINICAL TRIAL: NCT03780946
Title: Magnetic Compressive Technique for Pancreatic Intestinal Anastomosis
Acronym: MCTPIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2015-001-3
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Neoplasms; Pancreatitis, Chronic
Keywords: magnamosis; magnetic anastomosis; pancreaticojejunostomy
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Magnetic group: Magnetic anastomosis for pancreaticojejunostomy
  Interventions: Procedure: Magnetic anastomosis for pancreaticojejunostomy
- Control group: Traditional hand-sewn for pancreaticojejunostomy
  Interventions: Procedure: Traditional hand-sewn anastomosis

INTERVENTIONS:
Procedure: Magnetic anastomosis for pancreaticojejunostomy — Magnetic anastomosis for pancreaticojejunostomy
  Groups: Magnetic group
Procedure: Traditional hand-sewn anastomosis — Traditional manual anastomosis for pancreaticojejunostomy
  Groups: Control group

SUMMARY:
In recent five years, the investigators have successfully developed different types of magnets and utilized in biliojejunostomy, concomitant biliojejunostomy and pancreaticojejunostomy during Whipple. This study is designed as a prospective study by utilization of the bar-like magnets for pancreaticojejunostomy.

DETAILED DESCRIPTION:
Magnetic anastomosis has been attempted in continuous connection between bowel and bowel, vessels and vessels, biliary and gastrointestinal tracts, as well as in recanalization of the biliary stricture, and bilioenteric anastomotic stricture. During the past 15 years, the investigators have designed different types of magnets, and attempted these magnets in vascular, intestine, and biliary anastomosis in preclinical studies. In recent five years, we have successfully developed different types of magnets and utilized in biliojejunostomy, concomitant biliojejunostomy and pancreaticojejunostomy during Whipple. This study is designed as a prospective study by utilization of the bar-like magnets for pancreaticojejunostomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic neoplasm who needs pancreatic head resection, or central pancreatectomy or partial pancreatectomy, and then pancreaticojejunostomy
* Patients with dilated pancreatic duct secondary to chronic pancreatitis who needs Frey's procedure
* Patients with pancreatic injury who needs pancreatic head resection, or central pancreatectomy or partial pancreatectomy, and then pancreaticojejunostomy

Exclusion Criteria:

* Woman during pregnancy or lactation or anyone with mental disorder
* The wall of pancreatic incision is too thick so that the attractive force of magnetic device cannot meet the requirements of compression
* Any foreign body has been implanted in body, such as heart pacemaker.
* Surgical contraindication, including Child-Pugh C with hepatic encephalopathy, and anyone with heart, lung, kidney dysfunction or other organ dysfunction, and cannot tolerate surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with pancreatic neoplasm who needs pancreatic head resection, or central pancreatectomy or partial pancreatectomy, and then pancreaticojejunostomy.
  2. Patients with dilated pancreatic duct secondary to chronic pancreatitis who needs Frey's procedure.
  3. Patients with pancreatic injury who needs pancreatic head resection, or central pancreatectomy or partial pancreatectomy, and then pancreaticojejunostomy.
  4. Patients who are willing to join this clinical trial and informed consent form voluntarily.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula | From date of surgery to one month postoperatively
  Leakage of pancreatic fistula, which is defined according to Clinically relevant Pancreatic fistula (PF) was defined by the International Study Group of Pancreatic Surgery in 2016: a drain output of any measurable volume of fluid with an amylase level >3 times the upper limit of institutional normal serum amylase activity.

SECONDARY OUTCOMES:
Anastomotic stricture | one year from the date of surgery
  Anastomotic stricture, which will be verified by imaging studies or endoscopic investigations
Discharge of the magnets | 3 months from the date of surgery
  X-ray plain film is performed regularly to check the movement and discharge of the magnets

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China